CLINICAL TRIAL: NCT03494166
Title: Post-chemotherapy Symptom Management: Testing Intervention Sequences in a SMART Design
Brief Title: Post-chemotherapy Symptom Management SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Michigan State University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1711069340; R01CA225615 (NIH)
Record Dates: First submitted 2018-03-30; First posted 2018-04-11 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Chemotherapy, symptom management
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Following baseline, symptom management need (high versus low need) will be determined. The low need group will not receive interventions, but will be followed at week 4 for a brief symptom assessment and at week 13. The high need group will be randomly assigned to either: 1) SMSH alone or 2) TIP-C+SMSH for 8 weeks followed by continued 4 weeks of SMSH alone. We will mail the SMSH, printed in the survivor's preferred language, following randomization. All high need participants will receive weekly telephone contacts during weeks 1-12 to assess symptoms, deliver the assigned intervention, and assess intervention enactment and fidelity. After the initial 4 weeks, responders on depression will continue with the SMSH only. Non-responders will re-randomized to either continue with the SMSH alone or add TIP-C. Those initially randomized to TIP-C+SMSH will not be re-randomized. Total duration of each of the three intervention sequences is 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: Data collectors will be blinded to the arm of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Need Benchmark or Follow-up (No Intervention): In the low need benchmark or follow-up group, survivors completed detailed baseline and 13-week assessments (about 30-40 minutes) over the telephone. A brief assessment (about 5 minutes) at week 4 over the telephone was used to assess symptoms.
- High Need A: Start with SMSH alone for 4 weeks (Experimental): Participants were mailed the printed Symptom Management and Survivorship Handbook (SMH). The Group A participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMH to relieve symptoms. After 4 weeks, participants were re-randomized to continue in SMH for 8 more weeks or to add Telephone Interpersonal Counseling (TIPC) Intervention for the subsequent 8 weeks. If the TIPC was added, the counselor called the participant once per week for about 35-40 minutes to assess and discuss interpersonal relationships, communication, social support, managing symptoms and survivorship. At week 13, the participant completed the second assessment.
  Interventions: Behavioral: Start with SMSH alone
- High Need B: Start with SMSH+TIPC (Experimental): Participants were called every week for the first 8 weeks using a combination of TIP-C and SMH. The counselor called to assess and discuss interpersonal relationships, communication, social support, managing symptoms and survivorship. At the end of 8 weeks, the final 4 calls followed the SMSH alone protocol. At week 13, the second assessment was conducted.
  Interventions: Behavioral: Start with SMSH+TIPC

INTERVENTIONS:
Behavioral: Start with SMSH+TIPC — See arm/group descriptions
  Arms: High Need B: Start with SMSH+TIPC
Behavioral: Start with SMSH alone — See arm/group descriptions
  Arms: High Need A: Start with SMSH alone for 4 weeks

SUMMARY:
Survivors of solid tumors (N=451) who completed curative intent chemotherapy for a solid tumor within the past 2 years were interviewed at baseline and stratified as high or low need for symptom management based on comorbidity and depressive symptoms.

High need survivors were randomized initially to the 12-week Symptom Management and Survivorship Handbook (SMSH, N=282) or 12-week SMSH Telephone Interpersonal Counseling (TIPC, N=93) added during weeks 1-8. After 4 weeks of the SMSH alone, non-responders on depression were re-randomized to continue with SMSH alone (N=30) or add TIPC (N=31).

DETAILED DESCRIPTION:
Nearly 15.5 million Americans have survived cancer and virtually all have experienced symptoms from cancer treatment. Numerous symptom management interventions have been tested during active treatment, yet few have addressed the continuing fatigue, pain, depression, etc. that endure following the end of treatment.

Existing post-treatment symptom management research has targeted survivors months after the end of active treatment, overlooking the immediate post-treatment period. During this period, some survivors have their symptoms resolve naturally (low need for intervention), while others suffer from high symptom burden (high need for intervention), with 30% experiencing depression. Sample: Survivors of solid tumors (N=451) who completed curative intent chemotherapy for a solid tumor within the past 2 years.

Design: The SMART design incorporates two interventions with proven efficacy and addresses heterogeneity of survivors' responses by following the clinical logic of starting with one intervention, assessing its success, and continuing it when effective. High need survivors will be initially randomized to receive 1) weekly symptom assessment with referral for elevated symptoms to a printed Symptom Management and Survivorship Handbook (SMSH) or 2) a more intensive intervention adding Telephone Interpersonal Counselling (TIPC) to the SMSH. After 4 weeks, non-responders to SMSH alone on depression were re-randomized to continue SMSH for 8 more weeks to allow for symptom resolution, or TIPC added for the remaining 8 weeks.

The primary outcome was symptom severity index, secondary outcome was depressive symptoms. The hypotheses tests included comparisons of primary and secondary outcomes according tp first randomization and second randomization for non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Survivors must have a new diagnosis or localized recurrence of solid tumor cancer
* Be finishing curative intent adjuvant chemotherapy or chemoradiation, and do not have any subsequent cancer treatments planned, except for radiation therapy, hormonal therapy or trastuzumab for breast cancer.
* 18 years of age or older
* Have access to a telephone
* Understand English or Spanish
* Are not currently receiving counseling and/or psychotherapy

Exclusion Criteria:

* Diagnosis of a psychotic disorder in medical record verified by the recruiter
* Nursing home resident
* Bedridden
* Currently receiving counseling and/or psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Badger, PhD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Cancer Center at St. Joseph's, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: Yes
We will share the findings and data with other researchers, the public, and key stakeholders based on the principles that NIH has articulated regarding the sharing of study results and resources. The University of Arizona agrees that data sharing is essential for expedited translation of research results into knowledge, products, and procedures to improve health.
  Sharing of study results Manuscript based on results from the proposed study will be published in peer-reviewed journals. We will select "open access" options for these manuscripts whenever possible.
  Data Sharing Data from this study will be available to other researchers under the following conditions: 1) appropriate human subjects protection is in place; 2) data have been de-identified; and 3) study investigators have publicly presented and published key findings. Data and safety monitoring plan is described under Human Subjects.
Supporting Information: Study Protocol, SAP
Time Frame: Anticipate later part of 2022
Access Criteria: Data Sharing Data from this study will be available to other researchers under the following conditions: 1) appropriate human subjects protection is in place; 2) data have been de-identified; and 3) study investigators have publicly presented and published key findings. Data and safety monitoring plan is described under Human Subjects.

REFERENCES:
- [Result] Sikorskii A, Badger T, Segrin C, Crane TE, Chalasani P, Arslan W, Hadeed M, Morrill KE, Given C. A Sequential Multiple Assignment Randomized Trial of Symptom Management After Chemotherapy. J Pain Symptom Manage. 2023 Jun;65(6):541-552.e2. doi: 10.1016/j.jpainsymman.2023.02.005. Epub 2023 Feb 17. PMID 36801353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer survivors were recruited at a comprehensive cancer center, a federally qualified health center, and community settings in the Southwestern United States. Participants were informed they would be 1) randomized to SMSH or TIPC+SMSH and may be rerandomized after 4 weeks to continue with SMSH alone or add TIPC; 2) telephone assessment and intervention sessions were weekly for 13 weeks; 3) interventions were designed to help reduce symptoms and there were study incentives.
Pre-assignment Details: Of 500 consented individuals, 451 had a baseline interview, 71 were low need, 375 were high need and entered into randomization. Five participants were found ineligible. Three participants in the high need group dropped out after baseline before the first randomization. Three participants in the low need group were misclassified initially as high need and were randomized, resulting in 375 randomized and 68 continuing as low need without interventions.
Groups:
- Low Need Benchmark or Follow-up: In the low need benchmark or follow-up group, participants received baseline and 13-week assessments (about 30-40 minutes) over the telephone. A brief assessment (about 5 minutes) was done at week 4 over the telephone to assess symptoms. Approximately 35% of all participants were in this group.
- High Need- SMSH Alone for 4 Weeks, Depression Responders Continued With SMSH Alone for Weeks 5-12: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The High Need group participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. After 4 weeks, depression responders in the High Need group continued with the SMSH alone for weeks 5-12. Depression responders were survivors who started at severe at onset and ended at moderate or mild at a given time point (e.g., week 4), and survivors who started at moderate and ended at mild. At week 13, the participant was called to complete the second assessment.
- High Need-SMSH Alone for 4 Weeks, Depression Non-responders Continued With SMSH Alone for Weeks 5-12: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The High Need group participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. After 4 weeks, depression non-responders were re-randomized to either continue with the SMSH alone for weeks 5-12 or add Telephone Interpersonal Counseling (TIPC) to test the value added by the more intensive intervention. Symptom cases that remained moderate or became severe at week 4 are classified as non-responders. At week 13, the participant was called to complete the second assessment.
- High Need- SMSH Alone for 4 Weeks, Depression Non-responders Continued With SMSH+TIPC for Weeks 5-12: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The High Need group participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. After 4 weeks, depression non-responders were re-randomized to either continue with the SMSH alone for weeks 5-12 or add Telephone Interpersonal Counseling (TIPC) to test the value added by the more intensive intervention. The TIPC counselor assessed and discussed interpersonal relationships, communication, social support, managing symptoms, and survivorship. Symptom cases that remained moderate or became severe at week 4 are classified as non-responders. At week 13, the participant was called to complete the second assessment.
- High Need- SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The High Need group participant was called every week for the first 8 weeks using a combination of Telephone Interpersonal Counseling (TIPC) and SMSH. The TIPC counselor assessed and discussed interpersonal relationships, communication, social support, managing symptoms, and survivorship as well as asked about symptoms and suggest strategies from the SMSH to relieve symptoms. At weeks 9-12, the participant received the SMSH alone. At week 13, the participant was called to complete the second assessment.
- Drop-outs From SMSH Alone Prior to Week 4: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The High Need group participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. These participants were lost to attrition prior to the week 4 assessment for response or non-response.
Period: Overall Study
Arm/Group | Low Need Benchmark or Follow-up | High Need- SMSH Alone for 4 Weeks, Depression Responders Continued With SMSH Alone for Weeks 5-12 | High Need-SMSH Alone for 4 Weeks, Depression Non-responders Continued With SMSH Alone for Weeks 5-12 | High Need- SMSH Alone for 4 Weeks, Depression Non-responders Continued With SMSH+TIPC for Weeks 5-12 | High Need- SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12 | Drop-outs From SMSH Alone Prior to Week 4
Started | 71 | 204 | 30 | 31 | 93 | 17
Completed | 58 | 195 | 28 | 23 | 72 | 0
Not Completed | 13 | 9 | 2 | 8 | 21 | 17
Not completed — Death | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Lost to Follow-up | 2 | 2 | 2 | 2 | 14 | 0
Not completed — Withdrawal by Subject | 10 | 7 | 0 | 5 | 3 | 17
Not completed — Screen failure | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of 500 individuals who consented, 451 completed a baseline and 5 were ineligible.
Groups:
- High Need-SMSH Alone for 4 Weeks, Depression Responders Continued With SMSH Alone for Weeks 5-12: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The High Need group participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. After 4 weeks, depression responders in the High Need group continued with the SMSH alone for weeks 5-12. Depression responders are survivors who started at severe at onset and ended at moderate or mild at a given time point (e.g., week 4), and survivors who started at moderate and ended at mild. At week 13, the participant was called to complete the second assessment.
- Total: Total of all reporting groups
Arm/Group | Low Need Benchmark or Follow-up | High Need-SMSH Alone for 4 Weeks, Depression Responders Continued With SMSH Alone for Weeks 5-12 | High Need-SMSH Alone for 4 Weeks, Depression Non-responders Continued With SMSH Alone for Weeks 5-12 | High Need- SMSH Alone for 4 Weeks, Depression Non-responders Continued With SMSH+TIPC for Weeks 5-12 | High Need- SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12 | Drop-outs From SMSH Alone Prior to Week 4 | Total
Number analyzed (Participants) | 71 | 204 | 30 | 31 | 93 | 17 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.56 (13.13) | 58.76 (12.31) | 60.63 (12.88) | 53.83 (15.31) | 58.26 (12.93) | 60.18 (9.04) | 57.67 (12.73)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 22 | 32 | 4 | 6 | 14 | 2 | 80
  Female | 49 | 172 | 25 | 25 | 78 | 15 | 364
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Asian | 1 | 0 | 0 | 2 | 3 | 2 | 8
  Black or African American | 3 | 0 | 0 | 1 | 2 | 0 | 6
  White | 36 | 121 | 19 | 14 | 56 | 11 | 257
  More than one race | 1 | 0 | 0 | 2 | 3 | 0 | 6
  Unknown or not reported | 30 | 83 | 10 | 12 | 28 | 4 | 167
  Hispanic or Latino | 39 | 92 | 13 | 13 | 45 | 8 | 210
  Not Hispanic or Latino | 32 | 111 | 17 | 18 | 48 | 9 | 235
  Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 1
Symptom Severity [Mean (Standard Deviation); unit: units on a scale] — Symptoms were measured using the modified General Symptom Distress Scale (GSDS) assessment of 18 symptoms: fatigue, sleep difficulties, pain, headache, difficulty concentrating, lack of appetite, nausea, vomiting, constipation, diarrhea, numbness or tingling, skin rashes or sores, swelling, weakness, shortness of breath, cough, depression, and anxiety. Respondents indicated the severity of each symptom (0= not present,10= worst possible). A summed symptom severity index for 17 symptoms other than depression was derived. The potential range is 0-170, higher score reflects worse outcome.
  units on a scale | 24.70 (20.35) | 36.32 (25.48) | 46.97 (22.81) | 48.13 (26.46) | 37.28 (24.65) | 56.06 (34.18) | 36.96 (24.85)
Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Measured using Center for Epidemiological Studies-Depression (CES-D) 20-item scale. Potential score range is 0-60. Higher scores indicated worse outcome (higher depressive symptoms).
  units on a scale | 6.01 (4.66) | 13.01 (11.08) | 23.35 (12.69) | 23.72 (2.72) | 16.36 (13.42) | 19.25 (13.72) | 14.28 (11.92)

OUTCOME MEASURES:

1. Primary Outcome: Symptom Severity Index- Comparison of Two Groups Created by First Randomization
Description: Symptoms were measured using the modified General Symptom Distress Scale (GSDS) allowing for a quick assessment of 18 symptoms: fatigue, sleep difficulties, pain, headache, difficulty concentrating, lack of appetite, nausea, vomiting, constipation, diarrhea, numbness or tingling, skin rashes or sores, swelling, weakness, shortness of breath, cough, depression, and anxiety. Respondents indicated the severity of each symptom (0 = not present to 10 = worst possible). A summed symptom severity index for 17 symptoms other than depression was averaged over weeks 1-13 from each weekly contact, baseline, and 13-week interviews. Potential range 0-170, with higher score indicating worse outcome (greater severity). Because the collection of symptoms does not form a scale, internal consistency reliability was not applicable.
Time Frame: Weeks 1-13
Population: Of the 375 high-need survivors initially randomized, 282 received the Symptom Management and Survivorship Handbook (SMSH) alone and 93 received Telephone Interpersonal Counseling (TIPC) + SMSH.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- High Need A; Start With SMSH Alone: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The Group A participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. After 4 weeks, participants were re-randomized to continue in SMSH for 8 more weeks or to add Telephone Interpersonal Counseling (TIP-C) Intervention for the subsequent 8 weeks. If the TIP-C was added, the counselor called the participant once per week for about 35-40 minutes to assess and discuss strategies for managing symptoms, provide survivorship education, and discuss interpersonal relationships, communication, and social support. At week 13, the participant was called to complete the second assessment.
  Telephone Interpersonal Counseling (TIP-C): See arm/group descriptions
- High Need B: Start With SMSH+TIPC: Participant was called every week for the first 8 weeks using a combination of TIP-C and SMSH. The counselor assessed and discussed interpersonal relationships, communication, social support, managing symptoms, and survivorship. At the end of 8 weeks, the final 4 calls were focused on the SMSH protocol. At week 13, the second assessment was conducted.
  Telephone Interpersonal Counseling (TIP-C): See arm/group descriptions
Arm/Group | High Need A; Start With SMSH Alone | High Need B: Start With SMSH+TIPC
Number analyzed (Participants) | 282 | 93
score on a scale | 24.53 (0.68) | 25.86 (1.15)
Statistical Analysis 1: Comparison: High Need A; Start With SMSH Alone vs High Need B: Start With SMSH+TIPC; The null hypothesis was that the means in two arms were equal, the alternative hypothesis was that the means were not equal. We planned to randomize 224 survivors in approximately 3:1 ratio in the first randomization; power was 0.92 to detect the adjusted d=0.54 in the comparison of the SMSH and SMSH+TIPC in the first randomization. The planned number of 224 was exceeded because more survivors than planned were determined to have high need for symptom management; Test type: Superiority — Key parameter was the coefficient for the trial arm variable in the mixed model, reflecting average difference of group means over time (weeks 1-13); p = .31, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was set at .05; Linear mixed effects models were used for 13 repeated measures of symptom severity index, adjusting for baseline value; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-3.90 to 1.25], Standard Error of Mean 1.32 — The mean of the group that started with SMSH alone minus the mean of the group that started with SMSH+TIPC (average over time)

2. Primary Outcome: Symptom Severity Index- Comparison of Two Groups Created by Second Randomization
Description: Symptoms were measured using the modified General Symptom Distress Scale (GSDS) allowing for a quick assessment of 18 symptoms: fatigue, sleep difficulties, pain, headache, difficulty concentrating, lack of appetite, nausea, vomiting, constipation, diarrhea, numbness or tingling, skin rashes or sores, swelling, weakness, shortness of breath, cough, depression, and anxiety. Respondents indicated severity of each symptom (0 = not present to 10 = worst possible). A summed symptom severity index for 17 symptoms other than depression was averaged over weeks 5-13 from each weekly contact, baseline, and 13-week interviews. Potential range 0-170, higher value reflect worse outcome (greater symptom severity). Because the collection of symptoms does not form a scale, internal consistency reliability was not applicable.
Time Frame: Weeks 5-13
Population: Non-responders to the SMSH alone after 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Continue With SMSH Alone After Week 4: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). Participants were called weekly to ask about symptoms and suggest strategies from the SMSH to relieve symptoms.
- Add TIPC to SMSH After Week 4: Participant was called every week for 8 weeks using a combination of TIP-C and SMSH. The counselor assessed and discussed interpersonal relationships, communication, social support, managing symptoms, and survivorship.
  Telephone Interpersonal Counseling (TIP-C): See arm/group descriptions
Arm/Group | Continue With SMSH Alone After Week 4 | Add TIPC to SMSH After Week 4
Number analyzed (Participants) | 30 | 31
score on a scale | 35.94 (2.38) | 38.11 (2.49)
Statistical Analysis 1: Comparison: Continue With SMSH Alone After Week 4 vs Add TIPC to SMSH After Week 4; The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. The required sample size was 60 per group for .80 power or greater in two-tailed tests at the 0.05 level of significance using the effect size of Cohen's d=0.54 (adjusted for baseline and repeated measures). The actual sample size was smaller (61 total) due to the higher than planned rate of response to the SMSH alone by week 4; Test type: Superiority — The key parameter was the coefficient for the variable reflecting trial arm from the second randomization in the mixed model. This parameter reflected average difference between means of two groups over time (weeks 5-13); p = .52, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Linear mixed effects models were used for 9 repeated measures of symptom severity index (weeks 5-13), adjusting for baseline value; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-8.91 to 4.55], Standard Error of Mean 3.35 — The mean of the group that continued with SMSH alone minus the mean of the group that had TIPC added to the SMSH after week 4

3. Secondary Outcome: Depressive Symptoms- Comparison of Two Groups Created by First Randomization.
Description: Measured using Center for Epidemiological Studies-Depression (CES-D) 20-item scale. Potential score range is 0-60. Higher scores indicated worse outcome (higher depressive symptoms).
Time Frame: Week 13
Population: Of the 375 high-need survivors initially randomized, 282 started with the Symptom Management and Survivorship Handbook (SMSH) alone and 93 received Telephone Interpersonal Counseling (TIPC) + SMSH.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- High Need A-SMSH or TIP-C: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The Group A participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. After 4 weeks, participants were re-randomized to continue in SMSH for 8 more weeks or to add Telephone Interpersonal Counseling (TIP-C) Intervention for the subsequent 8 weeks. If the TIP-C was added, the counselor called the participant once per week for about 35-40 minutes to assess and discuss strategies for managing symptoms, provide survivorship education, and discuss interpersonal relationships, communication, and social support. At week 13, the participant was called to complete the second assessment.
  Telephone Interpersonal Counseling (TIP-C): See arm/group descriptions
- High Need B-TIP-C+SMSH: Participant was called every week for the first 8 weeks using a combination of TIP-C and SMSH. The counselor assessed and discussed interpersonal relationships, communication, social support, managing symptoms, and survivorship. At the end of 8 weeks, the final 4 calls were focused on the SMSH protocol. At week 13, the second assessment was conducted.
  Telephone Interpersonal Counseling (TIP-C): See arm/group descriptions
Arm/Group | High Need A-SMSH or TIP-C | High Need B-TIP-C+SMSH
Number analyzed (Participants) | 282 | 93
score on a scale | 11.89 (.55) | 12.30 (.99)
Statistical Analysis 1: Comparison: High Need A-SMSH or TIP-C vs High Need B-TIP-C+SMSH; The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. Sample size was determined by the power calculation for the primary outcome; Test type: Superiority — Key parameter was the coefficient for the trial arm from the first randomization variable in the linear regression model; p = .71, Regression, Linear — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Median Difference (Final Values) = -0.41, 95% CI 2-sided [-2.63 to 1.81], Standard Error of Mean 1.12 — The mean of group that started with SMSH alone minus the mean of the group that started with SMSH+TIPC

4. Secondary Outcome: Depressive Symptoms - Comparison of Two Groups Created by Second Randomization
Description: as for outcome 3
Time Frame: Week 13
Population: Non-responders to the SMSH alone after 4 weeks randomized for the second time (N=61).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Continue With SMSH Alone After Week 4 | Add TIPC to SMSH After Week 4
Number analyzed (Participants) | 30 | 31
score on a scale | 16.05 (1.93) | 16.81 (2.11)
Statistical Analysis 1: Comparison: Continue With SMSH Alone After Week 4 vs Add TIPC to SMSH After Week 4; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm from the second randomization variable in linear regression model; p = .79, Regression, Linear — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; The model included the adjustment for baseline value of the outcome; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-6.53 to 5.01], Standard Error of Mean 2.91 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events at baseline (week 0) and weekly for 13 weeks or up until their attrition date if applicable.
Description: Averse events/serious adverse events were identified during the implementation of the experimental protocols and were monitored by the Investigators in several ways: 1) Interviewers could identify both serious adverse events and/or adverse events during the completion of telephone interviews or telephone calls to schedule telephone interviews; 2) The interventionists could identify both serious adverse events and/or adverse events during their telephone contacts with the participants.
Groups:
- High Need A-SMH or TIP-C: Participants were mailed the printed Symptom Management and Survivorship Handbook (SMSH). The Group A participant was called every week for 4 weeks to ask about symptoms and suggest strategies from the SMSH to relieve symptoms. Calls were approximately 10 minutes. After 4 weeks, participants were re-randomized to continue in SMSH for 8 more weeks or to add Telephone Interpersonal Counseling (TIP-C) Intervention for the subsequent 8 weeks. If the TIP-C was added, the counselor called the participant once per week for about 35-40 minutes to assess and discuss strategies for managing symptoms, provide survivorship education, and discuss interpersonal relationships, communication, and social support. At week 13, the participant was called to complete the second assessment.
  Telephone Interpersonal Counseling (TIP-C): See arm/group descriptions
- High Need B-TIP-C+SMH: Participant was called every week for the first 8 weeks using a combination of TIP-C and SMSH. The counselor assessed and discussed interpersonal relationships, communication, social support, managing symptoms, and survivorship. At the end of 8 weeks, the final 4 calls were focused on the SMSH protocol. At week 13, the second assessment was conducted.
  Telephone Interpersonal Counseling (TIP-C): See arm/group descriptions
Arm/Group | Low Need Benchmark or Follow-up | High Need A-SMH or TIP-C | High Need B-TIP-C+SMH
All-Cause Mortality (participants affected / at risk) | 0/71 | 1/282 | 3/93
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/282 | 0/93
Other Adverse Events (participants affected / at risk) | 0/71 | 0/282 | 0/93

LIMITATIONS AND CAVEATS:
The larger than anticipated proportion of high need survivors resulted in a larger sample size for tests of hypotheses associated with first randomization. The higher than anticipated response rate to the SMSH at week 4 resulted in a lower number of survivors in the second randomization compared to the requirements of power analysis. On the other hand, a higher than anticipated rate of response to the SMSH alone led to a larger than planned number of responders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT03494166/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT03494166/ICF_000.pdf